CLINICAL TRIAL: NCT02380157
Title: Oral Potassium Supplementation in Healthy Men - Interactions With the Renin-angiotensin-aldosterone System and the Sympathetic Nervous System
Brief Title: Blood Pressure Regulation - Role of Potassium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Rasmus Dreier, Medical Doctor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: KARAASS-1
Record Dates: First submitted 2015-02-17; First posted 2015-03-05 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Blood Pressure; Hypertension
Keywords: Blood pressure; Potassium, Dietary; Renin-angiotensin-aldosterone system; Sympathetic nervous system
MeSH Terms: conditions — Hypertension | interventions — Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kaleorid (Experimental): 4 weeks treatment with Kaleorid, 750mg, 3 tablets 3 times daily.
  Interventions: Drug: Kaleorid, 750mg (trade name), Potassium chloride (active substance)
- Placebo (Placebo Comparator): 4 weeks treatment with Placebo tablets, 3 tablets 3 times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kaleorid, 750mg (trade name), Potassium chloride (active substance) — 4 weeks treatment with Kaleorid, 750mg, 3 tablets 3 times daily.
  Arms: Kaleorid
Drug: Placebo — 4 weeks treatment with Placebo tablets, 3 tablets 3 times daily.
  Arms: Placebo

SUMMARY:
Project titel: Oral potassium supplementation in healthy men - interactions with the renin-angiotensin-aldosterone system and the sympathetic nervous system Protocol number: KARAASS-1 EudraCT number: 2013-004460-66

Introduction The global burden of hypertension is huge. This project focuses on the role of potassium in human blood pressure regulation. A potassium rich diet lowers blood pressure and some studies have shown an increase in blood pressure during potassium depletion. Thus an inverse correlation between potassium intake and blood pressure exists. In this trial the objective is to test how an oral potassium supplementation, administered in form of the drug Kaleorid®, interacts with the renin-angiotensin-aldosterone system and the sympathetic nervous system.

Methods This is a randomized clinical placebo-controlled double-blinded crossover trial. A group of healthy men will be randomized to either 4 weeks treatment with the drug Kaleorid®, 750mg, 3 tablets 3 times daily or to 4 weeks treatment with placebo.

On day 26 in the first treatment period the participants meet at the hospital to start a 24-hours ambulatory blood pressure and collect a 48-hours urine sample. The same day a blood sample, an electrocardiogram (ECG) and a fat biopsy from the gluteal region will be done. The fat biopsy is expected to contain resistance vessels, which are to be investigated further in the laboratory.

On day 28 in the first treatment period the participants meet at the hospital again and are tested with an intravenous Angiotensin II infusion followed by continuous measurement of blood pressure and the following aldosterone response (using blood samples). Blood pressure will be measured with Finger Plethysmography and vascular tonus will be evaluated with the use of Impedance Cardiography, Finger Plethysmography and Doppler Ultrasound measurements of blood flow before, during and after the Angiotensin II infusion.

After this first period of treatment and testing a "washout" period of two weeks is inserted. After "washout", the participants crossover and starts the second treatment period.

Feasibility All necessary authorities have approved the trial and all cooperation is established.

DETAILED DESCRIPTION:
Project titel: Oral potassium supplementation in healthy men - interactions with the renin-angiotensin-aldosterone system and the sympathetic nervous system Protocol number: KARAASS-1 EudraCT number: 2013-004460-66

Objective

The objective of the study is to investigate how an oral potassium supplementation, administrated in form of the drug Kaleorid® regulates the human blood pressure. More specific the objective is to test how an oral potassium supplementation interacts with:

* The renin-angiotensin-aldosterone system and
* The sympathetic nervous system

To do this we plan to conduct a randomized clinical placebo-controlled double-blinded crossover trial to test how the drug Kaleorid® affects components in the renin-angiotensin-aldosterone system and the sympathetic nervous system compared with placebo in healthy men.

Background The global burden of hypertension is huge. The estimated number of adults with hypertension in the year 2000 was 972 million and this number is expected to increase by about 60% to a total number of 1.56 billion in 2025 worldwide (1). In Denmark, the estimated prevalence of hypertension among the adult population lies between 26% and 40% (2). Hypertension is thus a wide spread disease and it is further known, that hypertension is one of the most important modifiable risk factors for cardiovascular, cerebrovascular and renal disease (3;4). In this study we investigate the role of potassium in the regulation of the human blood pressure.

It is accepted knowledge, that a potassium rich diet lowers blood pressure as demonstrated in the well constructed DASH (Dietary Approaches to Stop Hypertension) study (5). In addition to a high potassium level the DASH diet also contained high levels of magnesium, calcium and low-fat dairy products and a low level of saturated fat, so whether the blood pressure lowering effect of the DASH diet was merely a result of the high potassium level or a result of the combined diet is difficult to tell. Nonetheless a meta-analysis demonstrated a significant systolic and diastolic blood pressure lowering effect of administration of an high-dose oral potassium supplementation compared to placebo or administration of an low-dose oral potassium supplementation (6). The risk of stroke, the main adverse outcome of long time hypertension, has also been demonstrated to be reduced with a high dietary potassium intake (7). And one study demonstrated that, the need for antihypertensive medication in hypertensive subjects can be reduced after an increase in the dietary potassium intake from natural foods (8). A high dietary potassium intake thus seems beneficial.

Furthermore potassium depletion seems to have the opposite effect of potassium supplementation. Both in normotensive men and in patients with essential hypertension the blood pressure increased during potassium depletion (9;10).

Taken together, there is reliable evidence for an inverse correlation between potassium intake and the level of blood pressure. Nevertheless the mechanism behind this apparent inverse correlation is still a conundrum. Different hypothesis has been developed, mostly on the basis of animal studies. In the rat kidney, potassium depletion is expected to elicit retention of sodium and thereby hypertension. At the level of the arterial wall potassium depletion is expected to lower the intracellular potassium level in smooth muscle cells, which would lead to a depolarization of the membrane and thereby elicit contraction, increased peripheral vascular resistance and hypertension. On the other hand a high potassium diet is expected to elicit an endothelium-dependent vasodilatation. Another postulated mechanism is that high potassium levels in the cerebrospinal fluid would decrease the sympathetic outflow from the brain and thereby blood pressure. The mentioned theories (11) are mainly based on animal studies.

It is known that a high potassium intake in humans results in an increased aldosterone level in the blood (12). The increased aldosterone level secures the body against hyperkalemia during potassium loading. In theory this rise in aldosterone should also elicit an inappropriate sodium and volume retention and thereby hypertension. But it does not. The blood pressure remains unchanged (12) or decreases after a rise in potassium intake.

So the question is - Why does the potassium stimulated aldosterone secretion not result in hypertension?

In the laboratory of Molecular Biology at the Department of Nephrology P, Rigshospitalet, we have found some interesting results regarding potassium and aldosterone. Working with an in vitro model of aldosterone secretion in the form of the human adrenocortical cell line H295R, which has been proven to be a model for studying the function of the human adrenal cortex (13;14), we found interactions between extracellular potassium and components of the renin-angiotensin-aldosterone system (RAAS). The H295R cell line is a model of the human adrenocortical zona glomerulosa cells, which normally are the site of synthesis and secretion of aldosterone in the human body. Aldosterone secretion from these cells is mainly stimulated by angiotensin II (Ang II), as part of the activation of the RAAS, and by extracellular potassium in situations with rising levels of extracellular potassium. These two secretagogues are traditionally being look upon as independent. But our studies showed interactions between the two systems. It was found that stimulation of the H295R cells with high levels of extracellular potassium decreased the amount of Ang II type 1 receptors in the membrane of the cells, measured as a fall in the specific binding of radioactive labelled Ang II to the cells (15). This reduction in specific binding of radioactive labelled Ang II, was followed by a potassium induced reduction in the expression of the Ang II type 1 receptor gene (AGTR1) (15). This means that the Ang II sensitivity of human aldosterone producing cells is reduced by high levels of extracellular potassium in vitro and the hypothesis is that high levels of extracellular potassium thus modulate the renin-angiotensin-aldosterone system.

Inspired by our results in the laboratory, the objective of this present study is to verify the existence of such inhibitory interactions between high potassium levels and RAAS in vivo. The overall purpose is to clarify the role of potassium in the regulation of human blood pressure.

Hypotheses In this trial 4 weeks treatment with the drug Kaleorid®, 750mg, 3 tablets 3 times daily, equivalent to 90 mmol potassium daily, is tested against 4 weeks treatment with placebo, 3 tablets 3 times daily in a crossover design. In the end of each treatment period tests are done to investigate components in the renin-angiotensin-aldosterone system and the sympathetic nervous system.

Primary hypothesis and primary endpoint:

The primary hypothesis is that treatment with Kaleorid® will reduce the Ang II sensitivity of the human adrenal cortex and thereby reduce the Ang II stimulated aldosterone secretion. This hypothesis will be tested with an intravenous Ang II infusion and measurement of the following aldosterone response in blood samples. The test will be done twice in each study participant, after treatment with Kaleorid® and after treatment with placebo.

Primary endpoint: Ang II stimulated S-aldosterone

Secondary hypothesis:

The secondary hypothesis is that treatment with Kaleorid® will also reduce the Ang II sensitivity of the smooth muscle cells in the human vascular resistance vessels through a down regulation of the Ang II receptors in the membrane of the smooth muscle cells. This would elicit vasodilatation and a fall in blood pressure To test this we will measure the blood pressure and evaluate vascular tonus before, during and after the above mentioned intravenous Ang II infusion. Blood pressure before, during and after the intravenous Ang II infusion will be measured with Finger Plethysmography and conventional brachial blood pressure measurement. Vascular tonus before, during and after the intravenous Ang II infusion will be evaluated with the use of Impedance Cardiography, Finger Plethysmography and Doppler Ultrasound measurements of blood flow. Impedance Cardiography and Finger Plethysmography will be used to estimate total peripheral resistance (TPR). Doppler Ultrasound will be used to measure blood flow and calculate resistance index (RI) in the renal artery, celiac artery and superior mesenteric artery.

Finally we will take a fat biopsy from the gluteal region of the study participants after each treatment period. In these biopsies we expect to find vascular resistance vessels, which we will investigate for receptorfunction and receptorexpression. Different receptors will be investigated, among them the Ang II type 1 receptor.

Tertiary hypothesis:

The tertiary hypothesis is that treatment with Kaleorid® will interact with activity in the sympathetic nervous system.

To test this potential interaction we plan to measure P-epinephrine and P-norepinephrine in blood and measure the content of epinephrine and norepinephrine in a urine sample at the end of each treatment period. We further plan to measure P-epinephrine and P-norepinephrine in blood before, during and after the above mentioned intravenous Ang II infusion.

Methods

Design:

This is a randomized clinical placebo-controlled double-blinded crossover trial designed to test how the drug Kaleorid® affects components in the renin-angiotensin-aldosterone system and the sympathetic nervous system compared with placebo in healthy men.

After inclusion and baseline screening a group of healthy men with a normal office blood pressure will be randomized to either 4 weeks treatment with the drug Kaleorid®, 750mg, 3 tablets 3 times daily or to 4 weeks treatment with placebo tablets, 3 tablets 3 times daily.

On day 26 in the first treatment period the study participants meet at the hospital and receive the equipment to measure a 24-hours ambulatory blood pressure and collect a 48-hours urine sample. On the same day a blood sample, an electrocardiogram (ECG) and a fat biopsy from the gluteal region will be done.

On day 28 in the first treatment period the study participants meet at the hospital again. This day to be further tested with the intravenous Ang II infusion followed by continuous measurement of blood pressure and the aldosterone response (using blood samples). Before, during and after the intravenous Ang II infusion blood pressure will be measured with Finger Plethysmography and conventional brachial blood pressure measurement. Vascular tonus before, during and after the intravenous Ang II infusion will be evaluated with the use of Impedance Cardiography, Finger Plethysmography and Doppler Ultrasound measurements of blood flow.

After this first period of treatment and testing a washout period of two weeks is inserted. After two weeks washout, the study participants crossover and starts the treatment again (second treatment period). The former Kaleorid® treated individuals become placebo treated individuals, and the former placebo treated individuals become Kaleorid® treated individuals. After another 4 weeks of treatment, the same tests as done after the first period of treatment is repeated.

Investigational drugs, Randomization, Blinding and Statistics:

The drug Kaleorid® and the placebo tablets constitute the investigational drugs in this clinical trial on humans. The drug Kaleorid® is purchased and delivered by the regional pharmacy of the Capital Region of Denmark. The placebo tablets are manufactured and delivered by the regional pharmacy of the Capital Region of Denmark. The same pharmacy is responsible for the randomization of the treatment, packing of the investigational drugs and labelling of the investigational drugs. The delivered tablet containers are not labelled with content, so the treatment is planned blinded for both study participants and investigators - so intentional double-blinded.

Since the design of the study is a cross-over design, statistics for paired data is planned to be used for evaluation of the results. A power calculation on the primary endpoint has been done according to standard criteria and 25 study participants are sufficient.

Experimental procedures:

Day 7 On day 7 in both treatment periods the study participants has a blood sample done to measure potassium, sodium, creatinine and eGFR. This is merely a safety blood sample to test that the study participants can tolerate the investigational drugs and do not develop hyperkalemia.

Day 26 On day 26 in both treatment periods the study participants meet at the hospital and receive the equipment to measure a 24-hours ambulatory blood pressure and collect a 48-hours urine sample. On the same day a blood sample, an electrocardiogram (ECG) and a fat biopsy from the gluteal region will be done.

The fat biopsies will be performed by a surgical skilled physician. After removal the biopsies are immediately transferred to ice-cold physiological buffer and transported to the laboratory at Glostrup Research Institute. At the laboratory small arterioles in the biopsies are dissected free from fat and connective tissue using a microscope. The dissected arterioles are sectioned into 1-2 mm length cylindrical segments which are either immediately used for vasomotor response studies or stored at -80°C for molecular studies. For vasomotor response studies, the isolated arteriole segments are mounted in a Mulvany-Halpern wire-myograph, whereby it is possible to test the physiological response of the vessel after adding different hormones e.g. Ang II. The molecular studies consist of quantitative real-time PCR to quantify the mRNA expression of the relevant receptor genes, western blot to analyse receptor protein expression and immunohistochemistry to analyse receptor localization.

Day 28 On day 28 in both treatment periods the study participants meet at the hospital again. After handing back the equipment used for the 24-hours ambulatory blood pressure and the urine sample the study participants are being tested with the intravenous Ang II infusion. The Ang II infusion is done with the study participant in a supine position. The Ang II infusion is given intravenously at a dosage of 5 ng/kg/min for 30 min. The chosen dosage and length of duration is based on other studies and is safe (16-18). Before, during and after the Ang II infusion blood samples are taking from another intravenous access to analyse the blood for S-aldosterone, P-angiotensin II, Plasma renin activity, P-epinephrine, P-norepinephrine and N-PRO-ANP.

Before, during and after the infusion the study participants are monitored closely. Blood pressure is measured with conventional brachial blood pressure measurement but also with Finger Plethysmography, which gives a continuous blood pressure assessment. Continuous Impedance Cardiography gives a continuous assessment of cardiac output and together with the blood pressure we are able to estimate total peripheral resistance during the Ang II infusion. In addition blood flow in the central arteries of the abdomen, are measured using Doppler Ultrasound.

Practical Feasibility This is a clinical trial with medicinal products in humans. The trial is approved by the Danish Health and Medicines Authority and the trial is registered in the EudraCT database with the EudraCT number: 2013-004460-66.

Under existing legislation clinical trials with medicinal products in humans must follow the rules of GCP (Good Clinical Practice). In accordance with this, the trial is monitored by the GCP unit at Copenhagen University Hospital.

The trial is approved by The Committees on Health Research Ethics in the Capital Region of Denmark.

In conclusion all necessary authorities have approved the trial.

Funding This study is supported by The Danish Heart Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 20-55
* Office Blood Pressure: < 140/90 mmHg
* BMI: 18,5-30,0 kg/m2
* Signed consent form

Exclusion Criteria:

* Diabetes mellitus
* Cerebrovascular disease, ischemic heart disease, peripheral artery disease
* Kidney disease
* Adrenal disease
* Ulcers
* Medical treatment
* Drug or alcohol abuse
* Pathological ECG
* Mental not suitable
* Hyperkalemia

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Angiotensin II stimulated S-aldosterone | Day 28 in each treatment period up to 70 days from start in the study

SECONDARY OUTCOMES:
Change in Angiotensin II stimulated blood pressure | Day 28 in each treatment period up to 70 days from start in the study
Change in Angiotensin II stimulated total peripheral resistance (TPR) | Day 28 in each treatment period up to 70 days from start in the study
Change in Angiotensin II stimulated resistance index (RI) in central vessels of the abdomen | Day 28 in each treatment period up to 70 days from start in the study
Level of receptor expression in resistance vessels from fat biopsies | Day 26 in each treatment period up to 70 days from start in the study
Level of receptor function in resistance vessels from fat biopsies | Day 26 in each treatment period up to 70 days from start in the study
P-epinephrine | Day 26 in each treatment period up to 70 days from start in the study
P-norepinephrine | Day 26 in each treatment period up to 70 days from start in the study
Urinary content of epinephrine | Day 26 in each treatment period up to 70 days from start in the study
Urinary content of norepinephrine | Day 26 in each treatment period up to 70 days from start in the study
Change in Angiotensin II stimulated P-epinephrine | Day 28 in each treatment period up to 70 days from start in the study
Change in Angiotensin II stimulated P-norepinephrine | Day 28 in each treatment period up to 70 days from start in the study

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Dreier, M.D., Principal Investigator — Department of Clinical Physiology and Nuclear Medicine, Glostrup Hospital, University of Copenhagen
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine, Glostrup Hospital, University of Copenhagen, Glostrup, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Ibsen H, Jorgensen T, Jensen GB, Jacobsen IA. [Hypertension--prevalence and treatment]. Ugeskr Laeger. 2009 Jun 8;171(24):1998-2000. Danish. PMID 19523360
- [Background] He J, Whelton PK. Epidemiology and prevention of hypertension. Med Clin North Am. 1997 Sep;81(5):1077-97. doi: 10.1016/s0025-7125(05)70568-x. PMID 9308599
- [Background] Whelton PK. Epidemiology of hypertension. Lancet. 1994 Jul 9;344(8915):101-6. doi: 10.1016/s0140-6736(94)91285-8. PMID 7912348
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Whelton PK, He J, Cutler JA, Brancati FL, Appel LJ, Follmann D, Klag MJ. Effects of oral potassium on blood pressure. Meta-analysis of randomized controlled clinical trials. JAMA. 1997 May 28;277(20):1624-32. doi: 10.1001/jama.1997.03540440058033. PMID 9168293
- [Background] Larsson SC, Orsini N, Wolk A. Dietary potassium intake and risk of stroke: a dose-response meta-analysis of prospective studies. Stroke. 2011 Oct;42(10):2746-50. doi: 10.1161/STROKEAHA.111.622142. Epub 2011 Jul 28. PMID 21799170
- [Background] Siani A, Strazzullo P, Giacco A, Pacioni D, Celentano E, Mancini M. Increasing the dietary potassium intake reduces the need for antihypertensive medication. Ann Intern Med. 1991 Nov 15;115(10):753-9. doi: 10.7326/0003-4819-115-10-753. PMID 1929022
- [Background] Krishna GG, Miller E, Kapoor S. Increased blood pressure during potassium depletion in normotensive men. N Engl J Med. 1989 May 4;320(18):1177-82. doi: 10.1056/NEJM198905043201804. PMID 2624617
- [Background] Krishna GG, Kapoor SC. Potassium depletion exacerbates essential hypertension. Ann Intern Med. 1991 Jul 15;115(2):77-83. doi: 10.7326/0003-4819-115-2-77. PMID 2058867
- [Background] Adrogue HJ, Madias NE. Sodium and potassium in the pathogenesis of hypertension. N Engl J Med. 2007 May 10;356(19):1966-78. doi: 10.1056/NEJMra064486. No abstract available. PMID 17494929
- [Background] Matthesen SK, Larsen T, Vase H, Lauridsen TG, Pedersen EB. Effect of potassium supplementation on renal tubular function, ambulatory blood pressure and pulse wave velocity in healthy humans. Scand J Clin Lab Invest. 2012 Feb;72(1):78-86. doi: 10.3109/00365513.2011.635216. Epub 2011 Dec 12. PMID 22149452
- [Background] Rainey WE, Bird IM, Mason JI. The NCI-H295 cell line: a pluripotent model for human adrenocortical studies. Mol Cell Endocrinol. 1994 Apr;100(1-2):45-50. doi: 10.1016/0303-7207(94)90277-1. PMID 8056157
- [Background] Rainey WE, Saner K, Schimmer BP. Adrenocortical cell lines. Mol Cell Endocrinol. 2004 Dec 30;228(1-2):23-38. doi: 10.1016/j.mce.2003.12.020. PMID 15541570
- [Background] 15. Egfjord M, Dreier R, Ravn L, Hofman-Bang J. Extracellular potassium modulated aldosterone secretion in relation to hypertensive states. 2013. Submitted.
- [Background] Bentley-Lewis R, Adler GK, Perlstein T, Seely EW, Hopkins PN, Williams GH, Garg R. Body mass index predicts aldosterone production in normotensive adults on a high-salt diet. J Clin Endocrinol Metab. 2007 Nov;92(11):4472-5. doi: 10.1210/jc.2007-1088. Epub 2007 Aug 28. PMID 17726083
- [Background] Cargill RI, Coutie WJ, Lipworth BJ. The effects of angiotensin II on circulating levels of natriuretic peptides. Br J Clin Pharmacol. 1994 Aug;38(2):139-42. doi: 10.1111/j.1365-2125.1994.tb04337.x. PMID 7981014
- [Background] Seidelin PH, McMurray JJ, Brown RA, Struthers AD. The effect of angiotensin II and noradrenaline alone and in combination on renal sodium excretion in man. Br J Clin Pharmacol. 1989 Jun;27(6):803-9. doi: 10.1111/j.1365-2125.1989.tb03443.x. PMID 2757896
- [Derived] Dreier R, Andersen UB, Forman JL, Sheykhzade M, Egfjord M, Jeppesen JL. Effect of Increased Potassium Intake on Adrenal Cortical and Cardiovascular Responses to Angiotensin II: A Randomized Crossover Study. J Am Heart Assoc. 2021 May 4;10(9):e018716. doi: 10.1161/JAHA.120.018716. Epub 2021 Apr 19. PMID 33870711